CLINICAL TRIAL: NCT04343755
Title: Phase IIa Study Exploring the Safety and Efficacy of Convalescent Plasma From Recovered COVID-19 Donors Collected by Plasmapheresis as Treatment for Hospitalized Subjects With COVID-19 Infection
Brief Title: Convalescent Plasma as Treatment for Hospitalized Subjects With COVID-19 Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of eligible patients due to change in standard therapy
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2020-0375
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
Keywords: Coronavirus; Covid19; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Convalescent Plasma (Experimental): Fresh or frozen plasma will be infused one time to patients
  Interventions: Biological: Convalescent Plasma

INTERVENTIONS:
Biological: Convalescent Plasma — Fresh or frozen plasma will be infused one time to hospitalized patients with COVID-19 infection

SUMMARY:
* This is a single arm phase IIa study of convalescent plasma for the treatment of individuals hospitalized with COVID-19 infection.
* Subjects will be considered as having completed the study after 60 (+/- 3) days, unless consent withdrawal or death occurs first.
* Interim analysis will be permitted as described in the statistical section 8.
* The final analysis will be conducted once the last subject completes the day 60 visit or withdraws from the study.

DETAILED DESCRIPTION:
Overall study design

* This is a single arm phase IIa study of convalescent plasma for the treatment of individuals hospitalized with COVID-19 infection.
* Subjects will be considered as having completed the study after 60 (+/- 3) days, unless consent withdrawal or death occurs first.
* Interim analysis will be permitted as described in the statistical section 8.
* The final analysis will be conducted once the last subject completes the day 60 visit or withdraws from the study.

Number of subjects

• Up to 36 patients in track 2, and 19 patients in track 3 as described in the statistical section 8.

Overall study duration

* The study begins when the first subject (this will likely be a donor) signs the informed consent. The study will end once the last enrolled subject completes the study (likely a recipient).
* The expected duration of the study is approximately 12 months.

ELIGIBILITY:
Donor Eligibility Criteria:

* Age 18-60
* A history of a positive nasopharyngeal swab for COVID-19 or a history of positive titer test.
* At least 14 days from resolution of COVID-19-associated symptoms including fevers
* One negative nasopharyngeal swabs for COVID-19 RNA
* Covid-19 neutralizing antibody >1:64
* Adequate venous access for apheresis
* Meets donor eligibility criteria in accordance to Hackensack University Medical Center (HUMC) Collection Facility at the John Theurer Cancer Center (JTCC) if collecting at the JTCC, and all regulatory agencies as describes in SOP 800 01 (Appendix A)
* Required testing of the donor and product must be performed in accordance to FDA regulations (21 CFR 610.40), and the donation must be found suitable (21 CFR 630.30)

Recipient Eligibility Criteria:

Recipients age >18 years old, are assigned to one of two clinical tracks, track 2 or 3, based on COVID-19 disease severity. Onset of first symptoms < 9 days.

Track 2:

* Hospitalized, moderate symptoms requiring medical care for COVID-19 infection
* Symptoms may include fever, dyspnea, dehydration among others
* Hypoxemia may be present but is not a requirement

Track 3:

* Requiring mechanical ventilation for the care of COVID-19 infection
* Requiring non-invasive positive pressure ventilation (NIPPV), such as continuous airway pressure (CPAP),bi-level positive airway pressure (BiPAP) or high flow nasal canula (HFNC).

Recipient exclusion criteria:

* History of severe transfusion reaction to plasma products
* Infusion of immune globulin within the previous 30 days
* AST or ALT > 10 x upper limit of normal
* Requirement for vasopressors
* COVID-19-associated acute kidney injury requiring dialysis
* DNR status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele L Donato, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Casadevall A, Scharff MD. Serum therapy revisited: animal models of infection and development of passive antibody therapy. Antimicrob Agents Chemother. 1994 Aug;38(8):1695-702. doi: 10.1128/AAC.38.8.1695. No abstract available. PMID 7985997
- [Background] Casadevall A, Scharff MD. Return to the past: the case for antibody-based therapies in infectious diseases. Clin Infect Dis. 1995 Jul;21(1):150-61. doi: 10.1093/clinids/21.1.150. PMID 7578724
- [Background] Casadevall A, Pirofski LA. Antibody-mediated regulation of cellular immunity and the inflammatory response. Trends Immunol. 2003 Sep;24(9):474-8. doi: 10.1016/s1471-4906(03)00228-x. No abstract available. PMID 12967670
- [Background] Casadevall A, Dadachova E, Pirofski LA. Passive antibody therapy for infectious diseases. Nat Rev Microbiol. 2004 Sep;2(9):695-703. doi: 10.1038/nrmicro974. PMID 15372080
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Background] Zhang JS, Chen JT, Liu YX, Zhang ZS, Gao H, Liu Y, Wang X, Ning Y, Liu YF, Gao Q, Xu JG, Qin C, Dong XP, Yin WD. A serological survey on neutralizing antibody titer of SARS convalescent sera. J Med Virol. 2005 Oct;77(2):147-50. doi: 10.1002/jmv.20431. PMID 16121363
- [Background] Sahr F, Ansumana R, Massaquoi TA, Idriss BR, Sesay FR, Lamin JM, Baker S, Nicol S, Conton B, Johnson W, Abiri OT, Kargbo O, Kamara P, Goba A, Russell JB, Gevao SM. Evaluation of convalescent whole blood for treating Ebola Virus Disease in Freetown, Sierra Leone. J Infect. 2017 Mar;74(3):302-309. doi: 10.1016/j.jinf.2016.11.009. Epub 2016 Nov 17. PMID 27867062
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Yeh KM, Chiueh TS, Siu LK, Lin JC, Chan PK, Peng MY, Wan HL, Chen JH, Hu BS, Perng CL, Lu JJ, Chang FY. Experience of using convalescent plasma for severe acute respiratory syndrome among healthcare workers in a Taiwan hospital. J Antimicrob Chemother. 2005 Nov;56(5):919-22. doi: 10.1093/jac/dki346. Epub 2005 Sep 23. PMID 16183666
- [Background] Ko JH, Seok H, Cho SY, Ha YE, Baek JY, Kim SH, Kim YJ, Park JK, Chung CR, Kang ES, Cho D, Muller MA, Drosten C, Kang CI, Chung DR, Song JH, Peck KR. Challenges of convalescent plasma infusion therapy in Middle East respiratory coronavirus infection: a single centre experience. Antivir Ther. 2018;23(7):617-622. doi: 10.3851/IMP3243. Epub 2018 Jun 20. PMID 29923831
- [Background] Arabi YM, Hajeer AH, Luke T, Raviprakash K, Balkhy H, Johani S, Al-Dawood A, Al-Qahtani S, Al-Omari A, Al-Hameed F, Hayden FG, Fowler R, Bouchama A, Shindo N, Al-Khairy K, Carson G, Taha Y, Sadat M, Alahmadi M. Feasibility of Using Convalescent Plasma Immunotherapy for MERS-CoV Infection, Saudi Arabia. Emerg Infect Dis. 2016 Sep;22(9):1554-61. doi: 10.3201/eid2209.151164. PMID 27532807
- [Background] Gunn BM, Yu WH, Karim MM, Brannan JM, Herbert AS, Wec AZ, Halfmann PJ, Fusco ML, Schendel SL, Gangavarapu K, Krause T, Qiu X, He S, Das J, Suscovich TJ, Lai J, Chandran K, Zeitlin L, Crowe JE Jr, Lauffenburger D, Kawaoka Y, Kobinger GP, Andersen KG, Dye JM, Saphire EO, Alter G. A Role for Fc Function in Therapeutic Monoclonal Antibody-Mediated Protection against Ebola Virus. Cell Host Microbe. 2018 Aug 8;24(2):221-233.e5. doi: 10.1016/j.chom.2018.07.009. PMID 30092199
- [Background] Wan Y, Shang J, Sun S, Tai W, Chen J, Geng Q, He L, Chen Y, Wu J, Shi Z, Zhou Y, Du L, Li F. Molecular Mechanism for Antibody-Dependent Enhancement of Coronavirus Entry. J Virol. 2020 Feb 14;94(5):e02015-19. doi: 10.1128/JVI.02015-19. Print 2020 Feb 14. PMID 31826992
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Crowe JE Jr, Firestone CY, Murphy BR. Passively acquired antibodies suppress humoral but not cell-mediated immunity in mice immunized with live attenuated respiratory syncytial virus vaccines. J Immunol. 2001 Oct 1;167(7):3910-8. doi: 10.4049/jimmunol.167.7.3910. PMID 11564809
- [Background] Tan M, Xiong X. Continuous and group sequential conditional probability ratio tests for phase II clinical trials. Stat Med. 1996 Oct 15;15(19):2037-51. doi: 10.1002/(SICI)1097-0258(19961015)15:193.0.CO;2-Z. PMID 8896138
- [Background] Tan MT, Xiong X. A flexible multi-stage design for phase II oncology trials. Pharm Stat. 2011 Jul-Aug;10(4):369-73. doi: 10.1002/pst.478. Epub 2010 Dec 8. PMID 22328328
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Convalescent Plasma
Started | 52
Completed | 40
Not Completed | 12
Not completed — Death | 11
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 13
Age, Continuous [Median (Full Range); unit: years] | 56 [27 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 30
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Hospitalized for COVID-19 But Not Intubated
Description: Mechanical ventilation rate at 7 days from starting treatment in hospitalized COVID-19 patients
Time Frame: 7 Days
Population: Of the 52 participants enrolled, 36 were not intubated at time of enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 36
Participants | 5

2. Primary Outcome: Primary Objective for Patients With COVID-19 Already Intubated
Description: Mortality rate at 30 days from starting treatment for patients with COVID-19
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 15
Participants | 7

3. Secondary Outcome: Duration of Hospitalization
Description: The duration of hospitalization is defined as the time in days from the first day of hospitalized to the date of discharge or death. Patients who are not discharged, are alive and still in the hospital on the date of closing follow-up, or lost follow-up on the date of closing follow-up will be considered censored on that date.
Time Frame: 60 Days
Population: The study was terminated early due to rapid change in standard therapy. This information was not collected or analyzed due to early termination.
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Mechanical Ventilation
Description: The duration of mechanical ventilation is defined as the time in days from the first day of using mechanical ventilation to the last day of using mechanical ventilation. All evaluable patients will be included and no censoring for this analysis.
Time Frame: 60 Days
Population: as for outcome 3
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Symptoms Resolution
Description: The time to symptom resolution is defined as the time in days from new therapy initiation to the first documented symptom resolution as assessed by local site. Patients whose symptom are not resolved, who are dead, or lost follow-up on the designed follow-up date will be censored on that date.
Time Frame: 60 Days
Population: Due to the early termination of the trial, data regarding this outcome were not collected.
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival
Description: Overall survival rate at 60 days from starting treatment for patients with COVID-19
Time Frame: 60 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 51
Participants | 40

7. Secondary Outcome: Rate of Virologic Clearance by Nasopharyngeal Swab at Day 10
Time Frame: 10 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 8
Participants | 7

8. Secondary Outcome: Rate of Virologic Clearance by Nasopharyngeal Swab at Day 30
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 8
Participants | 8

9. Secondary Outcome: Impact of Donor Titers Level on Efficacy
Time Frame: 60 Days
Population: as for outcome 3
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 0

10. Secondary Outcome: Impact of Donor Titers Level on Safety
Time Frame: 60 Days
Population: as for outcome 3
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 0

11. Secondary Outcome: Recipient Anti-SARS-CoV2 Titer Assessment on Days 0 (Pre-infusion)
Time Frame: 0 Days (pre-infusion)
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 51
Participants
  IgG Levels >=10,000 | 8
  IgG Levels 1000-10,000 | 23
  IgG Levels 500-1,000 | 4
  IgG Levels 100-500 | 8
  IgG Levels BLQ | 8

12. Secondary Outcome: Recipient Anti-SARS-CoV2 Titer Assessment on Days 3
Time Frame: 3 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 47
Participants
  IgG Levels >=10,000 | 23
  IgG Levels 1000-10,000 | 16
  IgG Levels 500-1,000 | 2
  IgG Levels 100-500 | 6
  IgG Levels BLQ | 0

13. Secondary Outcome: Recipient Anti-SARS-CoV2 Titer Assessment on Day 10
Time Frame: 10 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 47
Participants
  IgG Levels >=10,000 | 35
  IgG Levels 1000-10,000 | 7
  IgG Levels 500-1,000 | 0
  IgG Levels 100-500 | 4
  IgG Levels BLQ | 1

14. Secondary Outcome: Recipient Anti-SARS-CoV2 Titer Assessment on Day 30
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 33
Participants
  IgG Levels >=10,000 | 29
  IgG Levels 1000-10,000 | 3
  IgG Levels 500-1,000 | 0
  IgG Levels 100-500 | 1
  IgG Levels BLQ | 0

15. Secondary Outcome: Recipient Anti-SARS-CoV2 Titer Assessment on Day 60
Time Frame: 60 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 31
Participants
  IgG Levels >=10,000 | 25
  IgG Levels 1000-10,000 | 5
  IgG Levels 500-1,000 | 0
  IgG Levels 100-500 | 1
  IgG Levels BLQ | 0

ADVERSE EVENTS:
Time Frame: Safety assessment performed on post infusion day 0,3,10, 30, and 60 days
Arm/Group | Convalescent Plasma
All-Cause Mortality (participants affected / at risk) | 11/52
Serious Adverse Events (participants affected / at risk) | 24/52
Other Adverse Events (participants affected / at risk) | 0/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Convalescent Plasma (N=52)
Aneurysm (Investigations) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 1 (1)
Cerebral Edema (Nervous system disorders) | 1 (1)
Death (Infections and infestations) | 10 (10)
Readmission (Infections and infestations) | 2 (2)
Worsening Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Worsening Condition Intubation (Respiratory, thoracic and mediastinal disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT04343755/Prot_SAP_000.pdf